CLINICAL TRIAL: NCT06551740
Title: An Open-label, Randomized, Fed, Single-dose, 2-sequence, 2-period, Crossover Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of HUC2-344 and Co-administration of HUC2-344-R1 and HUC2-344-R2 in Healthy Volunteers
Brief Title: Phase 1 Study in Diabetes Mellitus(Fed)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUC2-344-1_FE
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Diabetes; Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- After a single dose of HUC2-344, co-administration of HUC2-344-R1 and HUC2-344-R2 (Experimental): Take 2 pills of comparative drugs first, and take 1 pill of IP after a 1 week of the break.
  Interventions: Drug: HUC2-344; Drug: HUC2-344-R1, HUC2-344-R2
- After co-administering HUC2-344-R1 and HUC2-344-R2 once, take single dose of HUC2-344 once. (Experimental): Take 1 pill of IP first, and take 2 pills of comparative drugs after a 1 week of the break.
  Interventions: Drug: HUC2-344; Drug: HUC2-344-R1, HUC2-344-R2

INTERVENTIONS:
Drug: HUC2-344 — per oral
Drug: HUC2-344-R1, HUC2-344-R2 — per oral

SUMMARY:
An open-label, randomized, Fed, single-dose, 2-sequence, 2-period, crossover phase 1 study in healthy volunteers.

DETAILED DESCRIPTION:
An Open-label, Randomized, Fed, Single-dose, 2-sequence, 2-period, Crossover Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of HUC2-344 and Co-administration of HUC2-344-R1 and HUC2-344-R2 in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged over 19 at screening
* Those whose BMI is between 18kg/m2 and 30kg/m2
* Those weight over 50kg(female 45kg)
* Those who are adequate to be subjects in this study upon judgment of the investigator after physical examination, clinical laboratory test, examination by interview, etc

Exclusion Criteria:

* Those who have clinically significant diseases or medical history below lists.

  1. Skin/mucous membranes
  2. Head and neck
  3. Eyes/appendages
  4. Ear, nose, and throat
  5. Thyroid/endocrine system
  6. Lungs/respiratory system
  7. Heart/circulatory system
  8. Abdomen/digestive system
  9. Kidney/urinary reproductive system
  10. Spine/musculoskeletal system
  11. Nervous/psychiatric system
  12. Blood/lymph/tumor
  13. Allergy/immune system
  14. Drug hypersensitivity
* Within 30 days prior to the first dose, the individual took medications significantly inducing or inhibiting drug-metabolizing enzymes such as barbiturates, or within 10 days prior to the first dose, took medications that could affect this study.
* Those who have participated in a bioequivalence study or other clinical trials and received investigational drugs within 6 months prior to the first dosing day.
* Within 8 weeks prior to the first dosing day, Those who have donated whole blood or within 2 weeks donated components, or received a blood transfusion within 4 weeks.
* Those who with a history of gastrointestinal resection surgery (excluding appendectomy or hernia repair) that could affect drug absorption, or those with gastrointestinal disorders.
* Within 1 month prior to the first dosing day, Those who meet the following conditions:

  1. For males, average alcohol consumption exceeding 21 drinks per week.
  2. For females, average alcohol consumption exceeding 14 drinks per week.
  3. Smoking more than an average of 20 cigarettes per day.
* Those who meet the following criteria:

  1. Known hypersensitivity reactions to active ingredients, excipients of investigational drugs, or non-quinolone drugs.
  2. Acute or chronic metabolic acidosis including type 1 diabetes mellitus, hyperglycemia, with or without ketoacidosis, or history of ketoacidosis.
  3. Estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73m² or severe and advanced renal impairment.
  4. End-stage renal disease or undergoing dialysis.
  5. Genetic issues such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
  6. Acute conditions affecting renal function such as dehydration, severe infection, cardiovascular collapse (shock), acute myocardial infarction, sepsis.
  7. Acute and unstable congestive heart failure.
  8. Receiving intravenous administration of iodinated contrast agents for radiographic studies.
  9. Diabetic ketoacidosis.
  10. Severe infections or severe systemic disorders.
  11. Malnutrition, starvation, cachexia, hypothalamic-pituitary dysfunction, or adrenal insufficiency.
  12. Acute or chronic conditions causing tissue hypoxia such as hepatic dysfunction, respiratory failure, acute myocardial infarction, shock, excessive alcohol consumption, dehydration, diarrhea, vomiting, or gastrointestinal disorders.
  13. Other reasons deemed unsuitable for participation in the clinical trial by the study investigator.
  14. For female subjects, pregnant, suspected pregnant, or lactating.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Cmax | 0,1,2,3,4, 4.5,5.5,6,7,8,9,10,12,24,48hours
  Maximum concentration of HUC2-344
Tmax | 0,1,2,3,4, 4.5,5.5,6,7,8,9,10,12,24,48hours
  Time of concentration
AUCt | 0,1,2,3,4, 4.5,5.5,6,7,8,9,10,12,24,48hours
  Area under the drug concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Seunghyeon Kang, Principal Investigator — H+YANGGI HOSPITAL
Locations (1):
- Huons, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided